CLINICAL TRIAL: NCT02413515
Title: Blood Pressure Control of Nifedipine GITS 60mg Treatment in Chinese Hypertensive Subjects Uncontrolled on Starting-dose Mono-therapy: A Prospective, Open-label, Multicenter, Single-arm, 8-week Study.
Brief Title: Blood Pressure Control of Nifedipine GITS 60mg Treatment in Chinese Hypertensive Subjects Uncontrolled on Starting-dose Mono-therapyo-therapy.
Acronym: ADEPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17677
Record Dates: First submitted 2015-04-02; First posted 2015-04-10 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Single arm study,the eligible subjects will receive Nifedipine GITS 60mg for 8 weeks
  Interventions: Drug: Nifedipine (Adalat GITS, BAY1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat GITS, BAY1040) — Nifedipine GITS 60 mg tablet, once daily, oral intake, for 8 weeks treatment

SUMMARY:
To evaluate antihypertensive efficacy and tolerability of Nifedipine GITS 60mg treated for 8 weeks in Chinese hypertensive subjects who failed to achieve BP control with the starting-dose antihypertensive monotherapy.

DETAILED DESCRIPTION:
Study design: it's a A prospective, open-label, multicenter, single-arm study. After a one- to two-week screening period, subjects receive Nifedipine GITS 60mg for 8 weeks.

The primary objective is to evaluate the antihypertensive efficacy of 8-week Nifedipine GITS 60mg treatment in Chinese hypertensive subjects who failed to achieve BP control with the starting-dose antihypertensive mono-therapy.

The secondary objective is to evaluate the tolerability of Nifedipine GITS 60mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to be included in the study only if they meet all of the following criteria:
* Aged 18 years or older, but less than 65 years;
* Either male or female
* BP is uncontrolled after at least 4 weeks of prior antihypertensive mono-therapy (the dosage of mono-therapy should be the starting dose of an angiotensin receptor blocker (ARB), angiotensin converting enzyme inhibitor (ACEI), b-blocker (BB), calcium channel blocker (CCB), or diuretic) both in the beginning and at the end of the screening period (uncontrolled BP is defined as MSSBP ≥140 and <160mmHg and/or MSDBP ≥ 90 and <100mmHg, and in the presence of diabetes mellitus: MSSBP ≥130 and <160mmHg and/or MSDBP ≥80 and <100mmHg);

Exclusion Criteria:

* Subjects meeting any of the following criteria are to be excluded from the study:
* Known hypersensitivity to nifedipine or to any of the following excipients, hypromellose, polyethylene oxide, magnesium stearate, sodium chloride, iron oxide red (E172/C.I.77491), cellulose acetate, polyethylene glycol 3350, hydroxypropyl cellulose, propylene glycol, titanium dioxide (E171/C.I.77891)
* Evidence of secondary hypertension such as coarctation of the aorta, pheochromocytoma, hyperaldosteronism, etc.

Severe gastro-intestinal tract narrowing; gastric banding; kock pouch (ileostomy after proctocolectomy)

* Evidence of cardiovascular shock
* Pregnant, possibly pregnant, planning to become pregnant or lactating women Received combination (two or more than two drugs combination) therapy or higher dosage (a higher dosage is defined as a higher dosage than the standard recommended starting dosage presented in the label of each drug) mono-therapy in the beginning or at the ending of the screening period.
* History of cerebrovascular ischemic event (stroke or transient ischemic attack [TIA]) within 6 months
* History of intracerebral hemorrhage or subarachnoid hemorrhage
* History of hypertensive retinopathy
* Any history of heart failure, New York Heart Association (NYHA) classification III or IV Severe coronary heart disease as manifested by a history of myocardial infarction or unstable angina in the past 12 months or a history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Clinically significant cardiac valvular disease
* History of arrhythmia
* Type 1 diabetes mellitus (DM)
* Hyperkalemia history: a serum potassium level above the upper limit of normal in the laboratory range;
* Liver disease or aspartate transaminase (AST) or alanine transaminase (ALT) levels >3 x upper limit of normal (ULN)
* Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) of <30 mL/min, or on hemodialysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with a Mean Sitting Systolic Blood Pressure (<130mmHg for subjects with diabetes and <140mmHg for others) of Nifedipine GITs 60mg | At week 8

SECONDARY OUTCOMES:
Changes in the Mean Sitting SBP(MSSBP) and Mean Sitting DBP(MSDBP) from baseline at Week 8 | baseline and week 8
Percentage of subjects with a Mean Sitting Systolic Blood Pressure Lower than 140mmHg and MSDBP less than 90 mmHg (130 and 80 for diabetis patients) of Nifedipine GITs 60mg | At week 2 and week 4
The percentage of subjects with a MSDBP lower than 90 (80 for diabetis) | At week 2 and week 4
The percentage of subjects achieving both a ≥10mmHg | At week 8
Time to reach the MSSBP target (based on the BP measurements during office visits) | up to week 8
  The MSSBP target means : 140 mmHg for others, 130 mmHg for diabetes
Changes in the 24-h, daytime (from 06:00 to 22:00), and nighttime (from 22:00 to 06:00) average SBP and DBP assessed by ABPM from baseline at Week 8 | baseline and week 8
incidence of all treatment-emergent adverse events | At week 8
incidence of drug-related treatment-emergent adverse events | at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- China (12):
  - Fuzhou, Fujian
  - Tangshan, Hebei
  - Wudan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Xi’an, Shanxi
  - Hangzhou, Zhejiang
  - Beijing
  - Shandong
  - Shanghai
  - Tangshang
  - Tianjin